CLINICAL TRIAL: NCT07138742
Title: Efficacy and Safety of Tacrolimus Eye Drops in Treatment of Vernal Keratoconjunctivitis
Brief Title: Tacrolimus Eye Drops in Treatment of Vernal Keratoconjunctivitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Ahmed Okasha, principle investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-7-5MD
Record Dates: First submitted 2025-08-08; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Vernal Keratoconjunctivitis
Keywords: vernal keratoconjunctivitis, Tacrolimus eye drops
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): This group will be treated by steroid eye drops
  Interventions: Drug: Steroid eye drops
- Intervention group 1 (Experimental): This group will be treated by compound Tacrolimus eye drop in 0.1% concentration
  Interventions: Drug: Tacrolimus eye drops
- Intervention group 2 (Experimental): This group will be treated by compound Tacrolimus eye drop in 0.01% concentration
  Interventions: Drug: Tacrolimus eye drops

INTERVENTIONS:
Drug: Steroid eye drops — steroid eye drops will be used in control group as usual regimen in treatment of vernal keratoconjunctivitis
  Arms: Control group
Drug: Tacrolimus eye drops — Compound Tacrolimus eye drops in 2 different concentrations will be assessed in treatment of vernal keratoconjunctivitis in terms of efficacy and safety being compared with steroid eye drops
  Arms: Intervention group 1; Intervention group 2

SUMMARY:
The purpose of the study is to evaluate efficacy and safety of topical Tacrolimus eye drops in different concentrations in treatment of vernal keratoconjunctivitis (VKC) comparing it with Steroid based usual topical regimen

DETAILED DESCRIPTION:
A hospital- based Prospective comparative randomized open label controlled trial . the study will be conducted on Patients with moderate to severe active VKC aged between (5-15) years old (pediatric age group). they will be divided into 2 groups control group will be treated with usual regimen ( steroid based) interventional group will be subdivided into 2 groups and each will be treated with Tacrolimus eye drops in 2 different concentrations

Follow up visits:

Will be scheduled 1st week , 2nd week then 4th week during the loading period Then every 2 weeks during the maintenance period Then monthly for another 3 months

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe active VKC aged between (5-15) years old (pediatric age group)

Exclusion Criteria:

1. Coexisting eye infections
2. Contact lens use
3. Systemic immunosuppressive drug use
4. Herpes keratitis
5. Recent ocular surgery or trauma
6. Known hypersensitivity to Tacrolimus
7. Ophthalmological comorbidities as cataract, glaucoma, and congenital eye anomalies
8. Impaired renal or hepatic functions

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Total subjective symptoms score (TSSS) | during loading period of drug intake ( 1 month )
  management of acute episodes : through Assessment of change in severity scores for symptoms and signs of inflammation from base line depending on Total subjective symptoms score (TSSS)
Total objective ocular signs score (TOSS) | during loading period of drug intake ( 1 month )
  management of acute episodes : through Assessment of change in severity scores for symptoms and signs of inflammation from base line depending on Total objective ocular signs score (TOSS)
visual acuity | during loading period of drug intake ( 1 month )
  management of acute episodes : with follow up of visual acuity using snellen chart
IOP measurement | during loading period of drug intake ( 1 month )
  management of acute episodes : with follow up IOP measurement in mmHg using applanation tonometry

SECONDARY OUTCOMES:
time of persistence | during maintenance period of drug intake ( 2 months)
  Reduction of exacerbations of inflammatory manifestations

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wan Q, Tang J, Han Y, Wang D, Ye H. Therapeutic Effect of 0.1% Tacrolimus Eye Drops in the Tarsal Form of Vernal Keratoconjunctivitis. Ophthalmic Res. 2018;59(3):126-134. doi: 10.1159/000478704. Epub 2017 Aug 12. PMID 28803239
- [Result] Zhao M, He F, Yang Y, Lin W, Qiu W, Meng Q, Zhang J, Zhou Z. Therapeutic efficacy of tacrolimus in vernal keratoconjunctivitis: a meta-analysis of randomised controlled trials. Eur J Hosp Pharm. 2022 May;29(3):129-133. doi: 10.1136/ejhpharm-2020-002447. Epub 2020 Nov 3. PMID 33144336
- [Result] Gokhale NS. Systematic approach to managing vernal keratoconjunctivitis in clinical practice: Severity grading system and a treatment algorithm. Indian J Ophthalmol. 2016 Feb;64(2):145-8. doi: 10.4103/0301-4738.179727. PMID 27050351